CLINICAL TRIAL: NCT04751799
Title: Impact of a VR Headset on Pain Perception and Satisfaction During Colposcopic Workup of Cervical Precancerous Lesions: a Multicenter Randomized-controlled Trial.
Brief Title: Virtual Reality: Influence on Satisfaction, Pain, and Anxiety in Patients Undergoing Colposcopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Günther Rezniczek, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VR-1
Record Dates: First submitted 2021-02-03; First posted 2021-02-12 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Cervical Dysplasia; Pain; Anxiety
Keywords: colposcopy; virtual reality; cervical dysplasia; pain; anxiety
MeSH Terms: conditions — Uterine Cervical Dysplasia; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective randomized open interventional study
Masking Description: No masking possible due to the nature of the intervention (using a virtual reality headset vs. not using a VR headset)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (no VR) (No Intervention): Patients undergoing colposcopy and colposcopically-guided biopsy without further intervention
- VR before and during colposcopy (Experimental): Patients undergoing colposcopy and colposcopically-guided biopsy with a VR headset for 15 minutes before colposcopy as well as during colposcopy.
  Interventions: Device: Virtual reality headset before colposcopy; Device: Virtual reality headset during colposcopy
- VR before colposcopy (Experimental): Patients undergoing colposcopy and colposcopically-guided biopsy with a VR headset for 15 minutes before colposcopy but not during colposcopy.
  Interventions: Device: Virtual reality headset before colposcopy

INTERVENTIONS:
Device: Virtual reality headset before colposcopy — Patients wear a virtual headset presenting 360° 3D views of relaxing environments
  Arms: VR before and during colposcopy; VR before colposcopy
Device: Virtual reality headset during colposcopy — Patients wear a virtual headset presenting 360° 3D views of distracting environments
  Arms: VR before and during colposcopy

SUMMARY:
Cervical cancer is one of the most common cancers in women and one of the leading causes of death in women worldwide. Pre-cancerous lesions (dysplasias) are detected by the screening smear test at the gynecologist's office and can thus contribute to a 100% chance of cure if they are clarified by a colposcopic examination as part of the dysplasia consultation.

To detect cervical dysplasia during colposcopic examination, the effect of diluted acetic acid on the epithelium of the cervix uteri is utilized. Metaplastic epithelium and low-grade dysplasia are visually noticeable by a slight white staining. Biopsies are then taken from these areas for further diagnosis.

The colposcopy itself and especially the colposcopic targeted biopsy of the cervix are painful. Virtual reality (VR) is a new method for 360° three-dimensional viewing of image content. A number of studies have shown that the use of VR can have a positive impact on the course of medical interventions. Randomized studies on the effectiveness of VR in a collective of women with colposcopically targeted biopsy of the cervix are not available according to a recent literature search (PubMed search of 12/30/2020; search terms: cervical biopsy, colposcopy, pain relief, pain control, virtual reality). In studies of our research group on colposcopy, we found increased pain scores especially in younger patients, but also in obese patients and smokers. A controlled study on the effectiveness of VR in colposcopically targeted biopsy is therefore useful.

In our study, we now want to answer the question under prospective conditions whether the use of VR before the start or before the start and during colposcopy compared to no intervention leads to a significant increase in patient satisfaction and/or a reduction in pain in the context of clarification colposcopy and colposcopically targeted biopsy.

DETAILED DESCRIPTION:
HPV and cervical cancer

Human papillomaviruses (HPV) are the most common sexually transmitted pathogens worldwide. The prevalence in the population is high. Epidemiological estimates suggest that 75-80% of sexually active adults acquire an HPV infection in the genital area at least once by the age of 50. However, up to 95% of these HPV infections are considered harmless and are spontaneously eliminated within 2 years in terms of immunological HPV clearance [1]. On the other hand, persistent infections with HPV of the high-risk group, e.g. HPV-16 and HPV-18, are the main cause for the development of cervical carcinoma and are also partly responsible for the development of vulvar carcinoma, vaginal carcinoma and anal carcinoma. HPV preferentially infects the epithelial cells of the anogenital region and, through incorporation of HPV DNA into the host genome and subsequent interference with the cell cycle control of the host cell, causes changes in the cervical epithelium that, if left untreated, may develop into precancerous lesions (so-called cervical intraepithelial neoplasia) and consecutively into invasive carcinoma of the cervix (cervical carcinoma). Specifically, the viral protooncogene E6 gene product couples to p53 and promotes its degradation, and the viral protooncogene E7 gene product forms a complex with the retinoblastoma gene product pRB and suppresses its tumor suppressor function [2]. Both the impairment of apoptosis and tumor suppressor function promote immortalization of infected basal cells in the transformation zone of the cervix uteri.

Cervical carcinoma is the third most common cancer in women worldwide, as well as the fourth leading cause of death in women worldwide. Cervical carcinoma accounted for 9% (n=529 800) of all new cancer cases and 8% (n=275 100) of cancer-related deaths in women in 2008 [3].

The precursor of cervical cancer is cervical intraepithelial neoplasia (CIN), which can lead to the development of squamous cell carcinoma (approximately 80% of all cervical cancers). Three grades of expression are distinguished in CIN (CIN1, CIN 2, and CIN 3). Compared with invasive cervical carcinoma, the occurrence of precancerous lesions of the cervix uteri is more widespread. It is estimated that approximately 100,000 women in Germany develop new dysplasias (CIN 1-3) annually, with a point prevalence of >200,000 [3, 4].

Colposcopy as a diagnostic method

Dysplasia of the cervix typically becomes conspicuous during the gynecological screening examination at the gynecologist. In this case, smears are taken from the ectocervix and endocervix and assessed by the cytologist after a Papanicolaou stain has been performed with regard to dysplastic cells and the quality of the smear. For further clarification of dysplastic changes, presentation to a specialized dysplasia consultation is recommended. During colposcopic examination, histological confirmation of dysplastic areas is performed by means of biopsy.

Colposcopy (visual examination of the vagina and the entrance to the uterus with optical magnification) is an integral part of early cervical cancer detection. It is used to visualize dysplastic areas on the cervix uteri and to determine their spatial expression. The magnifying glass allows a multilevel (3.5 to 30x) two-dimensional magnification. After visual identification of suspicious areas using 5% acetic acid (dysplasias become acetic white) and classification into "minor" (grade 1) or "major" (grade 2) changes according to the internationally used RIO classification, a targeted biopsy for exact determination of the degree of dysplasia is possible [4]. Only in this way is further individual therapy planning possible.

Pain sensation during colposcopic examination.

Colposcopy itself and especially colposcopic targeted biopsy of the cervix are painful [4, 5]. General practice is to use local analgesics, oral analgesics, or no analgesics during a colposcopically targeted biopsy of the cervix [5]. The use of nonpharmacologic methods to positively influence patient pain perception and satisfaction has been investigated in a number of studies. For example, in a prospective randomized study, our group demonstrated that classical music (Mozart, Symphony No. 40 in G minor, KV 550) [6] had no positive influence on satisfaction and pain perception. Similarly, in another randomized study, we found no positive influence on satisfaction and pain perception by using video colposcopy [7]. Virtual reality (VR) is a new method for 360° three-dimensional viewing of image content. A number of studies have shown that the use of VR can have a positive effect on the course of medical interventions. For example, in a systematic review and meta-analysis of 8 randomized trials with a total of 723 subjects, Ding et al showed lower postoperative pain scores after the application of VR in the context of various surgeries such as dental, knee, hemorrhoid surgery, and obstetric injury care [8].

Randomized trials of the effectiveness of VR in a collective of women undergoing colposcopy-targeted cervical biopsy are not available according to a recent literature search (PubMed search as of 12/30/2020; search terms: cervical biopsy, colposcopy, pain relief, pain control, virtual reality). In studies of our research group on colposcopy, we found increased pain scores especially in younger patients, but also in obese patients and smokers [7, 9]. Therefore, a controlled study on the effectiveness of VR in colposcopy-targeted biopsy is reasonable.

Aim of the study

Our study now aims to answer the question under prospective conditions whether the use of VR before initiation or before initiation and during colposcopy compared to no intervention leads to a significant increase in patient satisfaction and/or a reduction in pain in the context of clarification colposcopy and colposcopically targeted biopsy.

References

1. Workowski KA, Berman SM. Sexually transmitted diseases treatment guidelines, 2006. MMWR Recomm Rep. 2006;55:1-94.
2. Münger K, Scheffner M, Huibregtse JM, Howley PM. Interactions of HPV E6 and E7 oncoproteins with tumour suppressor gene products. Cancer Surv. 1992;12:197-217.
3. Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015;65:87-108. doi:10.3322/caac.21262.
4. Kühn W. Kolposkopie zur Früherkennung des Zervixkarzinoms. Pathologe. 2011;32:497-504. doi:10.1007/s00292-011-1480-9.
5. Heinrich J, Kühn W. Kolposkopie in Klinik und Praxis. 2nd ed. Berlin: De Gruyter; 2013.
6. Hilal Z, Alici F, Tempfer CB, Rath K, Nar K, Rezniczek GA. Mozart for Reducing Patient Anxiety During Colposcopy: A Randomized Controlled Trial. Obstet Gynecol. 2018;132:1047-55. doi:10.1097/AOG.0000000000002876.
7. Hilal Z, Alici F, Tempfer CB, Seebacher V, Rezniczek GA. Video Colposcopy for Reducing Patient Anxiety During Colposcopy: A Randomized Controlled Trial. Obstet Gynecol. 2017;130:411-9. doi:10.1097/AOG.0000000000002127.
8. Ding L, Hua H, Zhu H, Zhu S, Lu J, Zhao K, Xu Q. Effects of virtual reality on relieving postoperative pain in surgical patients: A systematic review and meta-analysis. Int J Surg. 2020;82:87-94. doi:10.1016/j.ijsu.2020.08.033.
9. Hilal Z, Rezniczek GA, Tettenborn Z, Hefler LA, Tempfer CB. Efficacy of Monsel Solution After Cervical Biopsy: A Randomized Trial. J Low Genit Tract Dis. 2016;20:312-6. doi:10.1097/LGT.0000000000000234.
10. Laux L, Glanzmann P, Schaffner P, Spielberger CD. Das State-Trait-Angstinventar (STAI). Theoretische Grundlagen und Handlungsanweisungen. Weinheim: Beltz; 1981.
11. Bornstein J, Bentley J, Bösze P, Girardi F, Haefner H, Menton M, et al. 2011 colposcopic terminology of the International Federation for Cervical Pathology and Colposcopy. Obstet Gynecol. 2012;120:166-72. doi:10.1097/AOG.0b013e318254f90c.
12. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009;42:377-81. doi:10.1016/j.jbi.2008.08.010.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Clinically indicated colposcopy in case of abnormal PAP smear for detection of precancerous lesions of the cervix uteri and/or clinical abnormality of the cervix uteri (e.g. leukoplakia) with biopsy

Exclusion Criteria:

* Eye diseases (e.g., glaucoma/cataracts) that impair viewing of VR content.
* Claustrophobia/agoraphobia or epilepsy
* Patients with insufficient knowledge of the German language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | immediately after procedure
  11-item VAS (0 = not satisfied at all, 10 = totally satisfied)

SECONDARY OUTCOMES:
Patient pain | during the colposcopy
  11-item VAS (0 = no pain, 10 = worst imaginable pain)
Patient pain | immediately after the colposcopy
  11-item VAS (0 = no pain, 10 = worst imaginable pain)
Patient anxiety | during the colposcopy
  11-item VAS (0 = not anxious at all, 10 = very anxious)
Surgical complications | 72 hours after colposcopy
  Questionnaire (mail-back or online) regarding pain, self-medicated pain medication, bleeding duration.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, Study Chair — Ruhr-Universität Bochum / Marien Hospital Herne
Locations (1):
- Marien Hospital Herne, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hecken JM, Halagiera P, Rehman S, Tempfer CB, Rezniczek GA. Virtual Reality for Anxiety Reduction in Women Undergoing Colposcopy: A Randomized Controlled Trial. J Low Genit Tract Dis. 2023 Jul 1;27(3):223-229. doi: 10.1097/LGT.0000000000000745. Epub 2023 May 11. PMID 37166026